CLINICAL TRIAL: NCT06195319
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Simufilam Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Simufilam Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTI-125-12
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Absorption; Metabolism; Excretion
MeSH Terms: interventions — Simufilam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Simufilam — 100 mg of [14C]-simufilam

SUMMARY:
To evaluate the absorption, metabolism, and excretion of [14C]-simufilam in healthy male subjects following a single oral administration of 100 mg of (approximately 100 µCi) [14C]-simufilam.

ELIGIBILITY:
Inclusion Criteria:

* Males of any race, between 18 and 55 years of age, inclusive.
* The subject has a body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive, and a total body weight between 50 and 110 kg, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination (at both screening and check-in), vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations (at both screening and check-in) as assessed by the Investigator (or designee).
* The subject is able to speak, read, and understand English and is willing to provide written informed consent.
* The subject is a non-smoker for the past 6 months.
* Must agree to use contraception History of a minimum of 1 bowel movement per day.
* The subject is willing and able to comply with all testing and requirements defined in the protocol.
* The subject must have completed a coronavirus disease (COVID-19) vaccine primary series ("fully vaccinate") at least 4 weeks prior to inpatient treatment day 1 of the study OR have COVID-19 virus serology consistent with prior vaccination or exposure.

Exclusion Criteria:

* The subject has had a clinically significant illness within 30 days prior to the Screening Visit.
* The subject has a significant history or clinical manifestation of any allergic, cardiovascular, dermatological, endocrine, gastrointestinal, hepatic, metabolic, neurological, psychiatric, pulmonary, renal, respiratory, or psychiatric disorder, as determined by the Investigator (or designee).
* The subject has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). A history of a cholecystectomy is exclusionary.
* Confirmed (e.g., 2 consecutive measurements) systolic blood pressure > 140 or < 90 mmHg, diastolic blood pressure > 90 or < 50 mmHg, and pulse rate > 100 or < 40 beats per minute. Minor deviations from the normal range may be allowed if deemed by the Investigator (or designee) to have no clinical significance.
* The subject has a clinically significant electrocardiogram (ECG) abnormality as evaluated by the Investigator (or designee).
* The subject has a clinically significant medical or laboratory abnormality or disease that, in the opinion of the investigator, should exclude the subject from the study, including:
* a. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or alkaline phosphatase (ALP) outside of the normal range at screening.
* Evidence of renal impairment (GFR < 90 mL/min/1.73m2 using the National Kidney Foundation CKD-EPI 2021 Creatinine Equation [9].
* Presence of congenital nonhemolytic hyperbilirubinemia (i.e., Gilbert's syndrome based on an assessment of total and direct bilirubin).
* The subject has a positive serum hepatitis B surface antigen test at the Screening Visit.
* The subject has or has had hepatitis C, as confirmed by a positive hepatitis C virus (HCV) antibody test at the Screening Visit.
* The subject has a positive human immunodeficiency virus (HIV) test at the Screening Visit
* The subject has been administered any vaccine in the 14-day period prior to dosing.
* The subject has used or intends to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 28 days prior to dosing, unless deemed acceptable by the Investigator (or designee) and Medical Monitor, in consultation with the Sponsor.
* The subject has used or intends to use any prescription medication within 14 days of dosing or over the counter (OTC) medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 48 hours of dosing and during the study unless deemed acceptable by both the Investigator (or designee) and Medical Monitor, in consultation with the Sponsor.
* The subject has used or intends to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the Investigator (or designee).
* The subject has received an investigational drug within 30 days prior to the Screening Visit.
* The subject has previously received simufilam.
* The subject has participated in ≥ 3 radiolabeled drug studies in the last 12 months (with most recent study to be at least 4 months prior to check-in to the study site where exposures are known to the investigator or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the investigator). The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States (US) Title 21 CFR 361.1.
* The subject has a history of substance abuse within 12 months of the Screening Visit or a current positive alcohol urine test or urine drug screen at the Screening Visit or at check-in.
* The subject has a history of regular alcohol consumption defined as greater than 14 drinks per week within six months prior to the Screening Visit. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits.
* The subject has used tobacco- or nicotine-containing products within 6 months prior to dosing or has a positive cotinine test at the Screening Visit or at check-in.
* The subject has consumed alcohol, caffeine, grapefruit, grapefruit juice, or xanthine-containing products within 72 hours before dosing or intends to use any of these products during the study.
* The subject has received blood products within 2 months prior to check-in.
* The subject has donated or lost a significant volume of blood (>500 mL) within a 90- day period prior to the Screening Visit or has donated plasma less than 2 weeks or platelets less than 6 weeks prior to the Screening Visit.
* The subject is unwilling to reside in the study unit for the duration of the study or unwilling to cooperate fully with the Investigator or site personnel.
* Subjects with poor peripheral venous access.
* Subjects with exposure to significant diagnostic or therapeutic radiation (e.g., serial x-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
AUC of total radioactivity, parent drug and metabolite(s) in plasma. | 10 days
  Area Under the Curve for each total radioactivity, parent drug and metabolite(s) in plasma.
Cmax of total reactivity, parent drug and metabolite(s) in plasma. | 10 Days
  Maximum concentration for each total radioactivity, parent drug and metabolite(s) in plasma.
Tmax of total reactivity, parent drug and metabolite(s) in plasma. | 10 Days
  Time to maximum concentration for each total radioactivity, parent drug and metabolite(s) in plasma.
Half-life of total reactivity, parent drug and metabolite(s) in plasma. | 10 Days
  Half-life for each total reactivity, parent drug and metabolite(s) in plasma.
Elimination rate constant of total reactivity, parent drug and metabolite(s) in plasma. | 10 Days
  Elimination rate constant for each total reactivity, parent drug and metabolite(s) in plasma.

SECONDARY OUTCOMES:
Percentage of total radioactivity recovered versus time. | 10 days
  Cumulative percentage of the administered radioactive dose recovered in urine, feces, and total excreta (urine and feces combined) versus time profiles.
Plasma and whole blood concentration of total radioactivity versus time. | 10 Days
  Plasma and whole blood concentration of total radioactivity versus time.
Plasma concentration of parent drug and metabolite(s) versus time. | 10 Days
  Plasma concentration of parent drug and metabolite(s) versus time.

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea, Madison, Wisconsin, United States